CLINICAL TRIAL: NCT04579133
Title: Phase II Randomized Study of Neoadjuvant Durvalumab (MEDI4736) Alone Versus Durvalumab (MEDI4736) With Olaparib (AZD2281) in Patients Ineligible for Cisplatin With Muscle-Invasive Urothelial Carcinoma of the Bladder Followed by Radical Cystectomy
Brief Title: Neoadjuvant Durvalumab Alone Versus Durvalumab With Olaparib in Patients Ineligible for Cisplatin With Muscle-Invasive Urothelial Carcinoma of the Bladder Followed by Radical Cystectomy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Not approved
Sponsor: Latin American Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LACOG 0219
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Bladder Cancer; Urothelial Carcinoma
Keywords: Bladder neoplasms; Bladder Cancer; Immunotherapy
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell | interventions — olaparib; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- durvalumab plus olaparib (Experimental): Durvalumab 1500 mg IV week 0, 3, 6 plus Olaparib tablets will be given orally on a continuous dosing schedule 300 mg BID OR 200 mg BID (if glomerular filtration rate [GFR] 31 to 50 mL/min) to complete 9 weeks of treatment.
  Interventions: Drug: Olaparib; Drug: Durvalumab
- durvalumab alone (Experimental): Durvalumab 1500 mg IV week 0, 3, 6 to complete 9 weeks of treatment
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Olaparib — 300 mg BID OR 200 mg BID (if glomerular filtration rate [GFR] 31 to 50 mL/min)
  Arms: durvalumab plus olaparib
Drug: Durvalumab — Durvalumab 1500 mg IV

SUMMARY:
This study is a phase II, randomized, open-label, clinical trial including patients with muscle-invasive transitional cell carcinoma of the bladder candidates for radical cystectomy. The study will include patients ineligible for cisplatin.

Patients will be centrally randomized in a 1:1 ratio to receive durvalumab plus olaparib (Arm A) or durvalumab alone (Arm B).

The clinical study´s hypothesis is that for patients with muscle-invasive transitional cell carcinoma of the bladder who are not fit for cisplatin-based neoadjuvant chemotherapy, Durvalumab monotherapy will have a similar efficacy to historical chemotherapy controls and Durvalumab in combination with olaparib will be associated with an even improved efficacy results in terms of pathologic complete response (pCR).

ELIGIBILITY:
Inclusion Criteria:

* 1. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

  2. Age > 18 years at time of study entry. 3. Evidence of muscle-invasive bladder cancer in a pretreatment transurethral biopsy sample.

  4. All histologic subtypes (with exception of small-cell carcinoma) will be eligible if urothelial carcinoma was the predominant histopathologic feature.

  5. Clinical stage T2-T4aN0M0 or T1-T4aN1M0 disease on imaging by American Joint Commission on Cancer, eighth edition.

  6. Available primary tumor tissue (formalin-fixed paraffin embedded FFPE or slides) from transurethral biopsy/resection for biorepository.

  7. Residual disease post transurethral resection prior to protocol inclusion and initiation.

  8. Patient must be planning to undergo a radical cystectomy at the time of randomization.

  9. Unfit for cisplatin-based neoadjuvant chemotherapy defined as the presence of at least one of the characteristics below:
  1. Creatinine clearance less than 60 mL/min;
  2. Grade 2 or worse hearing loss;
  3. Grade 2 or worse neuropathy;
  4. New York Heart Association class III heart failure. 10. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. 11. Body weight >30kg 12. Adequate normal organ and marrow function as defined below:
* Haemoglobin ≥10.0 g/dL with no blood transfusion in the past 28 days
* Absolute neutrophil count (ANC) 1.5 x 109/L
* Platelet count ≥100 x 109/L
* Total bilirubin ≤1.5 x institutional upper limit of normal (ULN).
* AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤5x ULN 13. Evidence of post-menopausal status or negative urinary or serum pregnancy test prior to ICF signature for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply: Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).

Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).

14. Female patients of childbearing potential who are not abstinent and intend to be sexually active with a non sterilized male partner must be in use of at least 1 highly effective method of contraception (see table in Section 7.1) before ICF signature/screening throughout the total duration of the drug treatment and the drug washout period (90 days after the last dose of durvalumab monotherapy). The study will not provide any method of contraception; this is responsibility of the patient in case of intention to participate in the study.

15. Male patients must use a condom during treatment and for 3 months after the last dose of study drug when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Female partners of male patients should also use a highly effective form of contraception. The study will not provide any method of contraception; this is responsibility of the patient in case of intention to participate in the study.

16. Patient is willing and able to comply with the protocol for the duration of the study, including undergoing treatment, scheduled visits, examinations and follow up.

Exclusion Criteria:

1. Participation in another clinical study with an investigational product during the last 3 weeks.
2. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
3. Any concurrent or within 3 weeks prior to study treatment systemic chemotherapy, IP, biologic, hormonal therapy or radiotherapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
4. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Patients must have recovered from any effects of any major surgery.
5. History of allogenic organ transplantation or double umbilical cord blood transplantation (dUCBT).
6. Patients with myelodysplastic syndrome/acute myeloid leukaemia or with features suggestive of MDS/AML
7. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

   1. Patients with vitiligo or alopecia
   2. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
   3. Any chronic skin condition that does not require systemic therapy
   4. Patients without active disease in the last 5 years may be included but only after consultation with the study physician
   5. Patients with celiac disease controlled by diet alone
8. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, uncontrolled cardiac arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
9. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
10. History of another primary malignancy except for

    1. Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence
    2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    3. Curatively treated in situ cancer of the cervix
    4. Ductal carcinoma in situ (DCIS) of the breast
    5. Stage 1, grade 1 endometrial carcinoma
11. Persistent toxicities (>Common Terminology Criteria for Adverse Event (CTCAE) grade 2) caused by previous cancer therapy, excluding alopecia
12. History of active primary immunodeficiency
13. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C (known positive HCV antibody) or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA. Screening for tuberculosis, hepatitis B, hepatitis C, and/or HIV infections is not required, unless there is clinical suspicion of these infections.
14. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

    1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
    2. Systemic corticosteroids at physiologic doses not to exceed <<10 mg/day>> of prednisone or its equivalent
    3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
15. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
16. Concomitant use of known strong CYP3A inhibitors (eg. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting study treatment is 2 weeks.
17. Concomitant use of known strong (eg. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort ) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting study treatment is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents
18. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy.
19. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
20. Prior randomisation or treatment in a previous durvalumab clinical study regardless of treatment arm assignment.
21. Patients who have received prior anti-PD-1, anti PD-L1, including durvalumab, or anti CTLA-4 antibodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Pathological complete response rate (pCR) | 24 weeks
  no evidence of invasive residual cancer (ypT0 or Tis/ypN0) in the surgical specimen.

SECONDARY OUTCOMES:
Overall Response rate (RR) | 9 weeks
  defined as proportion of patients with complete or partial response by RECIST v1.1.
Pathological Response including Downstaging to Non-muscle-invasive Cancer in the Surgical Specimen (pPR) | 24 weeks.
  defined as proportion of patients with pathological stage T1, Ta, and Tis.
Disease Free Survival (DFS) | 5 years.
  defined as time from randomization to disease recurrence or death, whichever occur first.
Overall Survival (OS) | 5 years.
  defined as time from randomization to death.
Safety (proportion of adverse events) | 24 weeks
  defined as proportion of patients with adverse events graded by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Pesquisa em Oncologia, Porto Alegre, Brazil